CLINICAL TRIAL: NCT00592904
Title: A Multi-Center, Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of E2007 (Perampanel) in Patients With Painful Diabetic Neuropathy (PDN) or Post-Herpetic Neuralgia (PHN)
Brief Title: Evaluating E2007 (Perampanel) in Patients With Painful Diabetic Neuropathy (PDN) or Post-Herpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-228; 2007-005495-13 (EudraCT Number)
Record Dates: First submitted 2008-01-03; First posted 2008-01-14 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-11

CONDITIONS: Neuralgia
Keywords: Neuralgia; neuropathy
MeSH Terms: conditions — Neuralgia | interventions — perampanel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007 — Perampanel doses will be up-titrated in 2 mg steps at minimum weekly intervals starting at 2 mg daily and up-titrated to 12 mg daily (taken orally).
  Other Names: Perampanel

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and continued efficacy of perampanel in patients previously enrolled in double-blind, placebo-controlled studies for Painful Diabetic Neuropathy (PDN) or Post-Herpetic Neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in this study:

1. Met and continues to meet all inclusion and none of the exclusion criteria for the preceding PDN or PHN study and received study drug or placebo under double-blind conditions.
2. Completed the preceding double-blind study End of Treatment (EOT) Visit no more than 12 weeks prior to Baseline (Visit 1) for the open-label study. The eligibility status of patients who do not enroll during this 12 week period will be evaluated on a case by case basis via discussion between the Investigator and the Sponsor.
3. Males and females ≥18 years of age. Female patients should be either of nonchildbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and practicing a medically acceptable method of contraception (e.g., abstinence, a barrier method plus spermicide, or intrauterine device [IUD]) for at least 1 month before the Baseline Visit (Visit 1) and for 1 month after the end of the study (Visit 16). They must also have a negative pregnancy test at Baseline (Visit 1). Female patients using hormonal contraceptives must also be using an additional approved method of contraception (e.g., a barrier method plus spermicide or IUD) throughout the study.
4. Provide written informed consent prior to entering the study and prior to undergoing any study-related procedures.
5. Is reliable, willing, and able to cooperate with the study procedures.

Exclusion Criteria:

Patients who meet the following criterion will be excluded from this study:

1. Patients who discontinued early for any reason from the preceding double-blind study.
2. Patients who have a clinically significant finding(s) that would make them unsuitable for the study in the opinion of the investigator or Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Laurenza, M. D., Study Director — Eisai Inc.
Locations (1):
- Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo: All subjects in this study received open-label perampanel, up-titrated in 2-mg increments from 2 mg/day to 12 mg/day. Subjects took 1 to 4 tablets orally once daily (QD), depending upon the subject's dose at that time. All subjects in this study previously completed a double-blind, placebo-controlled studies for PDN or PHN.
- PDN: Prior Treatment of Perampanel; Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo; PHN: Prior Treatment of Perampanel: All subjects in this study received open-label perampanel, up-titrated in 2-mg increments from 2 mg/day to 12 mg/day. Subjects took 1 to 4 tablets orally QD, depending upon the subject's dose at that time. All subjects in this study previously completed a double-blind, placebo-controlled studies for PDN or PHN.
Period: Overall Study
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel
Started | 57 | 148 | 27 | 30
Completed | 32 | 93 | 10 | 19
Not Completed | 25 | 55 | 17 | 11
Not completed — Adverse Event | 15 | 25 | 13 | 5
Not completed — Protocol Violation | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 16 | 1 | 2
Not completed — Lack of Efficacy | 2 | 7 | 2 | 3
Not completed — Physician Decision | 0 | 3 | 1 | 0
Not completed — Other | 3 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel | Total
Number analyzed (Participants) | 57 | 148 | 27 | 30 | 262
Age, Customized [Number; unit: Participants]
  <65 | 40 | 97 | 9 | 9 | 155
  ≥65 | 17 | 51 | 18 | 21 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 52 | 11 | 22 | 113
  Male | 29 | 96 | 16 | 8 | 149
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Asian | 2 | 1 | 0 | 0 | 3
    Black | 4 | 11 | 0 | 3 | 18
    White | 48 | 127 | 26 | 24 | 225
    Other | 3 | 9 | 1 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Short Form-McGill Pain Questionnaire (SF-MPQ): Sensory and Affective Scores, From Baseline to Week 48.
Description: Mean change from baseline to open-label study endpoint and other study visits in SF-MPQ scores sensory and affective). SF-MPQ was completed to assess intensity of pain over the past 48 days for all 15 descriptors: throbbing, shooting, stabbing, sharp, cramping, gnawing, hot-burning, aching, heavy, tender, splitting,tiring-exhausting, sickening, fear-causing, punishing-cruel. Each descriptor was scored by participant on a 4-point intensity scale (0=none to 3=severe) and totaled in each subclass (sensory range 0-45); higher scores indicated higher intensity of pain.
Time Frame: Baseline and Week 48
Population: Intent-to-Treat (ITT) Population: All enrolled subjects (starting at Visit 1) who took at least 1 dose of study drug and had at least 1 efficacy assessment in this trial comprised the ITT Population. All efficacy analyses were performed on the ITT Population. One subject had a protocol violation after consenting and was withdrawn from treatment.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel
Number analyzed (Participants) | 57 | 147 | 27 | 30
Scores on a Scale | -10.5 (8.41) | -8.1 (9.65) | -9.0 (6.72) | -9.8 (10.19)

2. Primary Outcome: Mean Change From Baseline in SF-MPQ Visual Analog Scale (VAS): From Baseline to Week 48.
Description: SF-MPQ VAS consists of a line 0 to 100 millimeters (mm) in length; range is 0 (no pain) to 100 mm (worst possible pain). Subjects placed a mark indicating the intensity of their pain. Distance from left-hand end of line was measured and entered on Case Report Form (CRF) as score in mm. Higher score indicates greater level of pain.
Time Frame: Baseline and Week 48
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel
Number analyzed (Participants) | 57 | 147 | 27 | 30
Scores on a Scale | -43.1 (23.17) | -33.7 (24.49) | -35.9 (24.55) | -35.4 (27.66)

3. Primary Outcome: Mean Change From Baseline in SF-MPQ Current Pain Intensity (CPI): From Baseline to Week 48
Description: Mean change from baseline in SF-MPQ (CPI) at study endpoint. Affective score ranges from 0-5. Higher scores indicate more severe pain (0=no pain, 1=mild, 2=discomforting, 3=distressing, 4=horrible, 5=excrutiating).
Time Frame: Baseline and Week 48
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel
Number analyzed (Participants) | 57 | 147 | 27 | 30
Scores on a Scale | -0.9 (0.71) | -1.0 (1.24) | -1.1 (0.57) | -1.3 (1.29)

4. Secondary Outcome: Analysis of Patient Global Impression of Change (PGIC) at Week 48/End of Treatment (EOT)
Description: The PGIC asked subjects to evaluate the change in their overall status compared with the start of open-label treatment on a scale ranging from 1 (very much improved) to 7 (very much worse). [Please note high withdrawl rate during study].
Time Frame: Baseline and Week 48
Population: Subset of ITT population used, including subjects that completed PGIC at Week 15 visit, and using BOCF (baseline observation carried forward) subjects that terminated prior to Week 15 received a 'No Change' if due to AE or Lack of Therapeutic Efficacy, subjects who discontinued due to other reasons used PGIC scores from Early Termination visit.
Measure: Number; unit: Participants
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel
Number analyzed (Participants) | 40 | 122 | 21 | 27
Participants
  Very much improved (1) | 8 | 22 | 5 | 6
  Much improved (2) | 16 | 33 | 3 | 9
  Minimally improved (3) | 12 | 39 | 4 | 7
  No change (4) | 3 | 13 | 3 | 5
  Minimally worse (5) | 0 | 12 | 2 | 0
  Much worse (6) | 1 | 2 | 3 | 0
  Very much worse (7) | 0 | 1 | 1 | 0

5. Secondary Outcome: Mean Change From Baseline in Short Form 36 Item (SF-36) Health Survey: Physical and Mental Component Scores From Baseline to Week 48/EOT
Description: Mean change from baseline in SF-36 Item Health Survey Scores at study endpoint. Each component on the SF-36 Item Health Survey is scored from 0-100 with higher scores reflecting better subject status.
Time Frame: Baseline and Week 48
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Painful Diabetic Neuropathy (PDN): Prior Treatment of Placebo | PDN: Prior Treatment of Perampanel | Post Herpetic Neuralgia (PHN): Prior Treatment of Placebo | PHN: Prior Treatment of Perampanel
Number analyzed (Participants) | 57 | 147 | 27 | 30
Scores on a Scale
  Physical Component Score | 5.48 (8.14) | 5.14 (9.36) | 1.72 (8.27) | 2.18 (9.30)
  Mental Component Score | 0.40 (8.90) | -2.32 (10.62) | -1.53 (10.77) | -3.12 (12.44)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) are those that started on or after first dose of open-label study drug up to and including 30 days after the last dose of open-label study drug.
Description: A subject who had the same TEAE more than once during the study was counted only once in the calculation of n (%) for that event.
Groups:
- Placebo: The participants who had previously received placebo during the double-blind study.
- Perampanel: The participants that had previously received perampanel during the double-blind study.
- Painful Diabetic Neuropathy: The participants that were being treated for PDN in the double-blind study and received either placebo or perampanel.
- Post Herpetic Neuralgia: The participants that were being treated for PHN in the double-blind study and received either placebo or perampanel.
Arm/Group | Placebo | Perampanel | Painful Diabetic Neuropathy | Post Herpetic Neuralgia
Serious Adverse Events (participants affected / at risk) | 11/84 | 25/178 | 31/205 | 5/57
Other Adverse Events (participants affected / at risk) | 72/84 | 132/178 | 160/205 | 44/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | Perampanel (N=178) | Painful Diabetic Neuropathy (N=205) | Post Herpetic Neuralgia (N=57)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 2 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Dementia (Nervous system disorders) | 1 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | Perampanel (N=178) | Painful Diabetic Neuropathy (N=205) | Post Herpetic Neuralgia (N=57)
Vertigo (Ear and labyrinth disorders) | 4 | 11 | 14 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 15 | 17 | 4
Nausea (Gastrointestinal disorders) | 6 | 6 | 11 | 1
Fatigue (General disorders) | 10 | 9 | 14 | 5
Gait disturbance (General disorders) | 6 | 9 | 12 | 3
Irritability (General disorders) | 5 | 4 | 7 | 2
Oedema peripheral (General disorders) | 5 | 13 | 16 | 2
Bronchitis (Infections and infestations) | 3 | 7 | 7 | 3
Nasopharyngitis (Infections and infestations) | 3 | 8 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 12 | 16 | 4
Contusion (Injury, poisoning and procedural complications) | 6 | 9 | 12 | 3
Fall (Injury, poisoning and procedural complications) | 10 | 15 | 21 | 4
Blood glucose increased (Investigations) | 5 | 2 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 13 | 14 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 11 | 12 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 5 | 3
Ataxia (Nervous system disorders) | 4 | 4 | 3 | 5
Balance disorder (Nervous system disorders) | 6 | 12 | 12 | 6
Dizziness (Nervous system disorders) | 36 | 63 | 76 | 23
Dysarthria (Nervous system disorders) | 7 | 9 | 12 | 4
Headache (Nervous system disorders) | 1 | 8 | 6 | 3
Somnolence (Nervous system disorders) | 15 | 35 | 38 | 12
Confusional state (Psychiatric disorders) | 4 | 5 | 4 | 5
Insomnia (Psychiatric disorders) | 1 | 6 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 4
Hypertension (Vascular disorders) | 5 | 7 | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No